CLINICAL TRIAL: NCT00102349
Title: HIV and HCV Intervention in Drug Treatment Settings
Brief Title: HIV and HCV Intervention In Drug Treatment Settings - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Robert Booth, Ph.D., University of Colorado at Denver
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Prevention
Other Study IDs: NIDA-CTN-0017-1
Record Dates: First submitted 2005-01-27; First posted 2005-01-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Behavior Therapy
Keywords: behavioral intervention
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to test two strategies to reduce the risk of contracting Human Immunodeficiency Virus (HIV) or Hepatitis C Virus (HCV) by reducing risk behaviors in patients undergoing drug detoxification.

ELIGIBILITY:
Volunteers will be IV drug users already enrolled in drug detoxification treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706
Dates: Start 2004-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
HIV/HCV injection risk behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Robert Booth, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (8):
- United States (8):
  - Denver Health & Hosp Authority, Denver, Colorado
  - Island Grove RTC, Greeley, Colorado
  - SSTAR (Stanley St. Treatment & Resources, Inc), Fall River, Massachusetts
  - James Gilmore Jr. Treatment Center, Kalamazoo, Michigan
  - Willamette Family Treatment Services, Eugene, Oregon
  - SSTAR of Rhode Island - North Kingstown, North Kingstown, Rhode Island
  - Recovery Center King Co.-Kent Detox, Kent, Washington
  - Recovery Center King Co.-Seattle Detox, Seattle, Washington